CLINICAL TRIAL: NCT01115010
Title: Effectiveness of a Proprietary Intraluminal Stiffening Wire in Decreasing Procedure Time and Improving Cecal Intubation Rate With Pre-owned Colonoscopes; a Randomized, Controlled Trial
Brief Title: Effectiveness of Stiffening Wire in Colonoscopy With Pre-Owned Colonoscopes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Colonoscope being used in study not repairable at economic cost.
Sponsor: Cornwall Regional Hospital (Other Government)
Collaborators: MoBay Hope Medical Center, Jamaica (Other)
Responsible Party: Jeffrey East, Cornwall Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: JE-1
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-07

CONDITIONS: Colonoscopy
Keywords: intubation rate; intubation time; stiffening device; stiffening wire

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stiffening wire only if difficulty (Experimental): Colonoscopy is performed with the unassisted colonoscope. The stiffening wire is introduced only if there is difficulty advancing the colonoscope and only after the tip has passed the splenic flexure. Difficulty is defined as failure to advance the tip of the scope after 5 minutes of trying.
  Interventions: Device: Colonoscope stiffening device
- Stiffening wire #1 transverse colon (Experimental): Colonoscopy is started with the unassisted colonoscope. Stiffening wire #1 is introduced on entry of the tip of the colonoscope into the transverse colon.
  Interventions: Device: Colonoscope stiffening device
- Stiffening wire #2 transverse colon (Experimental): Colonoscopy is started with the unassisted colonoscope. Stiffening wire #2 is introduced on entry of the tip of the colonoscope into the transverse colon.
  Interventions: Device: Colonoscope stiffening device

INTERVENTIONS:
Device: Colonoscope stiffening device — Colonoscopy is performed with the unassisted colonoscope (Olympus CF-100TL). The "standard" stiffening wire is introduced only if there is difficulty advancing the colonoscope and only after the tip has passed the splenic flexure. Difficulty is defined as failure to advance the tip of the scope after 5 minutes of trying. If difficulty is again encountered, the "firm" wire replaces the "standard" wire. Further difficulty requires removal of the firm wire and so on until cecal intubation is achieved or the procedure is abandoned.
  Other Names: ZUTR-141700 (Standard) and ZUTR-161700 (Firm) by Zutron Medical
  Arms: Stiffening wire only if difficulty
Device: Colonoscope stiffening device — "Standard" stiffening wire introduced routinely on entry into transverse colon. If difficulty is encountered (as defined previously), the "standard" wire is removed and attempts made to advance the colonoscope without it. Further difficulty requires introduction of the "firm" wire and so on until cecal intubation is achieved or the procedure is abandoned.
  Other Names: ZUTR-141700 (Standard) and ZUTR-161700 (Firm) by Zutron Medical
  Arms: Stiffening wire #1 transverse colon
Device: Colonoscope stiffening device — "Firm" stiffening wire introduced routinely on entry into transverse colon. If difficulty is encountered (as defined previously), the wire is removed and attempts made to advance the colonoscope without it. Further difficulty requires introduction of the "standard" wire and so on until cecal intubation is achieved or the procedure is abandoned.
  Other Names: ZUTR-141700 (Standard) and ZUTR-161700 (Firm) by Zutron Medical
  Arms: Stiffening wire #2 transverse colon

SUMMARY:
The study aims to determine whether a proprietary, FDA approved stiffening wire improves the efficiency of colonoscopy (that is, decreases the duration of the procedure) and/or enables complete visualization of the colon in a greater proportion of cases (than when the procedure is performed without it) with old, used colonoscopes.

Colonoscopes are designed with a delicate balance between stiffness and flexibility. Stiffness helps to prevent curling (looping) of the colonoscope in those sections of the colon that are not fixed to the wall of the abdominal cavity and flexibility enables successful negotiation of bends or flexures in the colon. As colonoscopes age, they lose stiffness and this makes it very challenging to advance the colonoscope all the way to the cecum (the upper end of the colon). Even when the cecum is successfully reached, it may take an inordinately long time.

In Jamaica, most endoscopists (General Surgeons and Gastroenterologists) use older, pre-owned colonoscopes imported from the USA, because the average patient and local health insurance companies cannot bear the level of fees that would enable cost recovery for new equipment.

The stiffening wires (in two grades of stiffness) used in this study are passed through the biopsy channel of the colonoscope only after its tip has passed the upper end of the descending colon and entered the transverse colon. The device is safe when used as recommended by the manufacturers (and approved by the FDA), and does not appear to increase risk over and above the risk of colonoscopy with the unassisted colonoscope. Although the device clearly improves the stiffness of the colonoscope, there is no research evidence that it actually works in practice, either to improve cecal intubation rate or to decrease procedure time. It is therefore also unclear whether the possible benefit of using the device is achieved if introduced at the first opportunity allowed by the manufacturers or only after difficulty is encountered with the unassisted colonoscope.

In this study, patients are randomly assigned to one of 3 "interventions". One group has colonoscopy performed with the colonoscope alone and the wires are only introduced if there is difficulty advancing the colonoscope after it has passed into the transverse colon ("difficulty" defined as failure to advance the tip of the colonoscope after 5 minutes). In the 2nd and 3rd groups, the assigned wire will be introduced as soon as the colonoscope enters the transverse colon and is removed if "difficulty" is encountered, as defined above. The different phases of colonoscopy will be timed with a stop watch and when a sufficient number of patients has been accrued, the investigator will be able to compare the time it takes to complete the procedure with and without the wires as well as the proportion of cases in which the cecum was reached with and without the assistance of the wires.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older having screening or diagnostic colonoscopy

Exclusion Criteria:

* Previous hysterectomy
* Previous radical prostatectomy
* Clinical presentation or imaging study suggesting presence of lesion that could obstruct passage of colonoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cecal intubation | 10 months

SECONDARY OUTCOMES:
Time to cecal intubation | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M East, MD, Principal Investigator — Cornwall Regional Hospital
Locations (1):
- Mobay Hope Medical Center, Montego Bay, Saint James Parish, Jamaica

REFERENCES:
- [Background] Odori T, Goto H, Arisawa T, Niwa Y, Ohmiya N, Hayakawa T. Clinical results and development of variable-stiffness video colonoscopes. Endoscopy. 2001 Jan;33(1):65-9. doi: 10.1055/s-2001-11174. PMID 11204990
- [Background] Shah SG, Saunders BP. Aids to insertion: magnetic imaging, variable stiffness, and overtubes. Gastrointest Endosc Clin N Am. 2005 Oct;15(4):673-86. doi: 10.1016/j.giec.2005.08.011. PMID 16278132
- [Background] Sivak MV. Gastroenterologic Endoscopy. Second Edition. W.B. Saunders, 1999.
- [Background] Zutron Medical. Colonoscope stiffening device. http://zutronmedical.storesecured.com/items/Endoscope-Stiffening-System/list.htm . 2009. Ref Type: Electronic Citation
- [Background] Smith PG, Morrow RH. Field Trials of Health Interventions in Developing Countries: A Toolbox. 2nd ed. London: Macmillan Education, 1996.
- [Background] Othman MO, Bradley AG, Choudhary A, Hoffman RM, Roy PK. Variable stiffness colonoscope versus regular adult colonoscope: meta-analysis of randomized controlled trials. Endoscopy. 2009 Jan;41(1):17-24. doi: 10.1055/s-0028-1103488. Epub 2009 Jan 21. PMID 19160154
- [Background] Baron TH. The variable stiffness colonoscope: a scope for all seasons? Am J Gastroenterol. 2002 Dec;97(12):2942-3. doi: 10.1111/j.1572-0241.2002.07091.x. No abstract available. PMID 12492173
- [Derived] East JM. Effect of a proprietary intraluminal stiffening wire device on cecal intubation time and rate with used colonoscopes; a randomized, controlled trial. BMC Res Notes. 2013 Feb 4;6:48. doi: 10.1186/1756-0500-6-48. PMID 23379922